CLINICAL TRIAL: NCT01043302
Title: Multicenter Cross Sectional Study of Primary Intestine Lymphoma: Treatment Outcome and Quality of Life
Brief Title: Multicenter Cross Sectional Study of Primary Intestine Lymphoma
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Kim, Seok Jin, Samsung Medical Center
Other Study IDs: 2008-09-060
Record Dates: First submitted 2010-01-04; First posted 2010-01-06 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-07

CONDITIONS: Non-Hodgkin Lymphoma of Intestine
Keywords: lymphoma, intestine, outcome, quality of life
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Surgery+chemotherapy: Primary mass was resected and systemic chemotherapy was performed as an adjuvant treatment
- Chemotherapy: Only treated with chemotherapy

SUMMARY:
The purpose of this study is to determine whether whether surgical resection followed by chemotherapy is superior to systemic chemotherapy alone in terms of treatment outcome and quality of life (QOL) in patients with primary intestinal lymphoma.

DETAILED DESCRIPTION:
Intestine is the one of commonly involved extranodal sites of non-Hodgkin's lymphoma (NHL). Thus, small and large Intestine account for approximately 30-40% of primary gastrointestinal tract lymphoma. More than 70% of intestinal lymphoma presents as localized disease, and surgery such as bowel resection is performed in many patients with intestinal lymphoma for diagnosis and treatment. However, it is still unclear whether surgical resection followed by chemotherapy is superior to systemic chemotherapy alone in terms of treatment outcome and quality of life (QOL). Thus, we analyze the clinical features and treatment outcome of patients with NHL of intestine, and at the same time perform a multicenter cross-sectional study about the QOL in survivors of intestine NHL. We evaluates the treatment outcomes of patients with intestine NHL from hospitals affiliated with the Consortium for Improving Survival of Lymphoma (CISL) in Korea. We assess the QOL of survivors who completed their treatment using the EORTC QLQ-C30 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Primary intestine lymphoma.

Definition of primary intestine lymphoma:

1. Dominant site should be small and large intestine with or without regional lymph node involvement
2. Distant lymph node involvement can be allowed if the intestine lesion is the presenting site
3. Contiguous involvement of other organs such as liver, spleen can be allowed

Exclusion Criteria:

* Intestine involvement as a dissemination process in stage IV nodal lymphoma

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: University hosptial, general hospital, Cancer institute
Sampling Method: Probability Sample
Enrollment: 545 (Actual)
Dates: Start 2008-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Overall survival | Study entry

SECONDARY OUTCOMES:
Quality of life | Study entry

CONTACTS AND LOCATIONS:
Overall Officials: Seok Jin Kim, MD.,PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim SJ, Kang HJ, Kim JS, Oh SY, Choi CW, Lee SI, Won JH, Kim MK, Kwon JH, Mun YC, Kwak JY, Kwon JM, Hwang IG, Kim HJ, Park J, Oh S, Huh J, Ko YH, Suh C, Kim WS. Comparison of treatment strategies for patients with intestinal diffuse large B-cell lymphoma: surgical resection followed by chemotherapy versus chemotherapy alone. Blood. 2011 Feb 10;117(6):1958-65. doi: 10.1182/blood-2010-06-288480. Epub 2010 Dec 9. PMID 21148334